CLINICAL TRIAL: NCT02874469
Title: Impact of an Intensive Care Diary on Post-traumatic Stress Disorder on Patients After a Resuscitated Sudden Death and His Relatives
Brief Title: Impact of an Intensive Care Diary on Post-traumatic Stress Disorder After a Resuscitated Sudden Death
Acronym: COREABOR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Lille (Other)
Collaborators: Ministry of Health, France (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2014_06; 2014-A01213-44 (Other: ID-RCB number, ANSM)
Record Dates: First submitted 2016-08-17; First posted 2016-08-22 (Estimated); Last update posted 2025-12-16 (Actual); Status verified 2020-08

CONDITIONS: Sudden Death; Sudden Cardiac Arrest
Keywords: sudden death; post-traumatic stress disorder; psychological distress; diary; resuscitation
MeSH Terms: conditions — Death, Sudden; Death, Sudden, Cardiac; Stress Disorders, Post-Traumatic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (first period) (No Intervention): Patients treated as recommended with usual care in a center.
- Group with diary (second period) (Experimental): Intervention group = On top of usual care, an intensive care unit diary will be implemented for patients within the first 8 hours following their admission.
  Interventions: Other: Diary

INTERVENTIONS:
Other: Diary — The diary was specifically created for the purpose of the present study by personal working at ICU at CHRU of Lille (France).
  All relatives, doctors and paramedics close to the patient during his hospital stay are allowed to write some comments inside the diary when he is comatose.
  The diary will be implemented during the second period of the study within the first 8 hours after admission.
  It will be given to the patients themselves at discharge or to their relatives in case of in-hospital death. An anonymous copy will be kept by investigators.
  Arms: Group with diary (second period)

SUMMARY:
Sudden death is a public health problem with more than 300,000 cases per year in USA and 40,000 cases per year in France. Moreover, despite all recent therapeutic improvements (therapeutic hypothermia, new techniques of resuscitation…), the prognosis remains drastically poor and less than 50% of the patients admitted alive at hospital will survive to the event at 1 year.

Outside all medications and technical care to improve patient prognosis, a psychological evaluation looks also critical to detect the occurrence of a "post traumatic stress syndrome". In fact, along with the event severity, a variable period of amnesia related to coma may favor the occurrence of such a syndrome and psychological issues, which at the end may lead to impairment of patient quality of life.

Previous studies have evaluated the impact of an intensive care unit diary on psychological distress in patients and relatives in the context of severe traumatisms. Such an evaluation has however never been done in the specific setting of sudden death and the frequency of this syndrome is unknown in this context.

Aim The aim of the present study is to evaluate the impact of an intensive care unit diary on the occurrence of a "post traumatic stress syndrome" after a sudden death.

Secondary objectives

* To evaluate the frequency of the occurrence of a "post traumatic stress syndrome" and other psycho traumatic symptoms after sudden death
* To evaluate the impact of an intensive care unit diary on the severity of this syndrome, psycho traumatic symptoms, and psychopathologic comorbidities
* To evaluate the impact of the diary on psycho traumatic symptoms and their severity in patient's relatives
* To evaluate the satisfaction of the patients and their relatives regarding medical cares in both groups (with and without diary)
* Comparison of nurse diagnostic (psychological distress) and diagnostic made by dedicated personal with a specific formation in psychology
* Qualitative evaluation of the diary
* Evaluation of the paramedical feeling before and after the diary input in practice

DETAILED DESCRIPTION:
The COREABOR Study is an open label, prospective, that will compare patients with sudden death who will be included during 2 successive periods of time: first a period of control and then a period of intervention.

Interventional study.

Altogether, 330 patients with resuscitated sudden death will be screened during the whole study period allowing to include 96 patients in the study (alive at 3 months after the event, estimated survival rate of 30%). For each screened patient, 2 relatives will be selected to participate to the study (n=660).

To avoid biases, the control group of 48 patients will be included first and treated as recommended with usual care in center. Then, the 48 patients of the intervention group will be included during the second period of the study and the intensive care unit diary will be implemented only at this time.

In the intervention group (second period with diary), a maximal delay of 8 hours is allowed to implement the diary for each patient after admission in centre.

Visit 0 (V0): inclusion The study will recruit patients in the total incapacity to give their own consent for medical reasons (comatose patients) at admission. Subsequently a written inform consent of a relative will first be obtained and the patient's written consent will be obtained as soon as possible afterwards.

Period 1: control group Medical care as usually performed in center and as recommended.

Period 2: intervention group (intensive care unit diary) On top of usual care, an intensive care unit diary will be implemented for all patients within the first 8 hours following their admission. At discharge, the diary will be given to the patients themselves or to their relatives in case of in-hospital death. An anonymous copy will be kept by investigators.

For all patients A psychological evaluation will be performed at 1 month (V1), 3 months (V2) and 6 months by phone contact only (V3) using the following elements Auto-questioner (PDI) Nurse diagnosis Psychological evaluation by dedicated personal (CAPS and mini-DSMIV)

For relatives A psychological evaluation will be performed at 3 months (V2) and 6 months by phone contact only (V3)

ELIGIBILITY:
Inclusion criteria =

* Patients who experienced a sudden death and who are admitted alive in our center
* Patients who benefited from therapeutic hypothermia (and/or care to limit fever occurrence)

Relative's inclusion criteria :

* Relatives of a patient that fit inclusion/exclusion criteria

Exclusion Criteria =

Patient's non-inclusion criteria :

* Death or transfer in another center within the first 8 hours of admission in our center
* Pregnancy
* Patients who refuse to participate after being awake after initial coma

Relative's non-inclusion criteria :

* Relatives who refuse to participate after being awake after initial coma

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 173 (Actual)
Dates: Start 2014-12-31 (Actual); Primary Completion 2023-12 (Actual); Study Completion 2023-12 (Actual)

PRIMARY OUTCOMES:
Rate of occurrence of "post traumatic stress disorder" | 3 months
  Rate of occurrence of "post traumatic stress syndrome" (CAPS score over 39) at 3 months after resuscitation after sudden death

SECONDARY OUTCOMES:
Peritraumatic Distress Inventory (PDI) Scale | 1 month
  PDI is a scale of self-evaluation of 13 items to determine distress reactions emotional of a person at the time of a traumatic event and in the minutes and hours. People who have a high risk of distress Peritraumatic develop post-traumatic stress disorder.
Psychiatric comorbidities | 3 and 6 months
  Psychiatric comorbidities evaluated by the mini DSM IV (Diagnostic and Statistical Manual of Mental Disorders - IV) for patients
Rate of "Post traumatic stress disorder" for patients | 6 months
  Rate of "Post traumatic stress disorder" (CAPS score over 39) for patients
Rate of "Post traumatic stress disorder" for relatives | 3 and 6 months
  Rate of "Post traumatic stress disorder" (CAPS score over 39) for relatives
Nurse diagnosis | 3 months
  Comparison of nurse diagnosis and diagnosis made by dedicated personal with a specific formation in psychology
Qualitative evaluation of the diary | 6 months
  Qualitative evaluation of the diary by satisfaction questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Gilles LESMESLE, MD, PhD, Principal Investigator — University Hospital, Lille
Locations (1):
- Hôpital Cardiologique - USIC - CHRU, Lille, France

IPD SHARING:
Plan to Share IPD: No